CLINICAL TRIAL: NCT00831155
Title: Brain Substrates of Extinction Based Treatment for Nicotine Dependence
Brief Title: Extinction Based Treatment for Nicotine Dependence
Acronym: Extinction01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009639
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Nicotine Dependence
Keywords: smoking; nicotine patches; extinction based treatment
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Extinction Based Group (EBT): switch to smoking denicotinized cigarettes while wearing a 21mg/day nicotine patch for one month prior to their quit date.
  Interventions: Drug: Nicotine Patches, Denicotinized Cigarettes
- 2 (No Intervention): Nicotine Replacement Group (NRT): smoke their usual brand of cigarettes up to the quit date.

INTERVENTIONS:
Drug: Nicotine Patches, Denicotinized Cigarettes — Both groups will receive standard Nicotine Replacement Therapy after the quit date. The Extinction Based group will receive Nicotine patches and denicotinized cigarettes before their quit date
  Arms: 1

SUMMARY:
The purpose of this study is to test two quit smoking therapies and to study brain function while each therapy is being used. You will be randomly assigned (like flipping a coin) to one of the two groups. The first therapy is Extinction-Based therapy (EBT). If you are in this group, you will switch to smoking denicotinized cigarettes while wearing a 21 mg/d nicotine patch for one month prior to your quit date. The second therapy is a standard Nicotine Replacement therapy (NRT). If you are in this group, you will smoke your usual brand of cigarettes up to the quit date. Following the quit date, both groups will undergo standard nicotine replacement therapy (21 mg/d for 6 weeks; 14 mg/d for 2 weeks, 7 mg/d for 2 weeks).

In addition to the above, we will recruit a sample of former smokers who are now regular users of e-cigarettes. This group [ECIG] will undergo the same screening and baseline assessments as the EBT and NRT groups up to the completion of fMRI1.

DETAILED DESCRIPTION:
If you agree to be in this study, you will be asked to sign the consent form prior to any tests or procedures. You will be asked to come to the laboratory for a screening session. The screening session will take approximately 1.5 hours to complete, including all questionnaires, physical and sample collection. Pregnant or nursing mothers will not be allowed to participate in this study. If you test positive for illegal drug use, you will not be allowed to participate in this study. Depending on the results of the screening procedures you may not be eligible for the study. If you do not have any medical conditions that would make your participation risky, and you feel comfortable participating in the study, you will be given instructions regarding the rest of the study sessions and be asked to return.

Smoker participants who complete the screening visit (described above) and meet all study requirements will then complete 8 lab visits, 1 fMRI training session, 3 fMRI sessions, and 2 follow-up visits. ECIG participants who complete the screening visit and meet all study requirements will complete 1 fMRI training session and 1 fMRI session.

First you will be randomly assigned (like drawing out of a hat) to a study group, either the EBT or NRT group. In the extinction-based therapy (EBT) group, participants will switch to smoking denicotinized cigarettes while wearing a 21 mg/d nicotine patch for one month prior to their quit date; meanwhile, smokers assigned to the nicotine replacement therapy (NRT) group will smoke their usual brand of cigarettes up to the quit date. Following the quit date, both groups will undergo standard nicotine replacement therapy (21 mg/d for 6 weeks; 14 mg/d for 2 weeks, 7 mg/d for 2 weeks).

Eight lab visits (V1 - V8) will be conducted during the 16 weeks following enrollment in the study. These visits will be largely identical, except that instructions and reminders to you about upcoming events will vary from session to session. At each lab visit the following will be collected: vitals (heart rate, blood pressure and weight); breath CO (Carbon Monoxide) and saliva samples for testing smoking and nicotine levels; and measures of smoking withdrawal and mood. You will be given daily diaries to record your smoking behavior and study medication. You will be given instructions on how and when to use all study materials. Advice on quitting and minimal support will be provided as requested at these visits. Each lab visit will require 20-30 minutes of your time.

Directly following V1 you will undergo a training session, during which you will be familiarized with all aspects of the fMRI sessions including tasks and equipment. You will be situated in a scanner simulator, which simulates the sounds and equipment used in the fMRI scanner.

One task will require you to view pictures of people smoking and people doing everyday activities. After the task, you will be quizzed on the pictures you saw. During another task, you will be presented with a stream of gray, yellow, or blue colored circles and instructed to press a button every time you see a "Go" trial while inhibiting a response (not pressing the button) when you are presented with a "No-Go" trial. The training session will require 1 hour of participant time.

fMRI Sessions:

You will be asked to complete three fMRI scanning sessions: a baseline scan (fMRI-1); a scan 4 weeks after you start treatment (fMRI-2); and a final scan 24 hours after your quit date (fMRI-3). The first 20 minutes of each scanning session will follow the same protocol as a lab visit. Following this, for fMRI-1 and fMRI-2 you will be asked to smoke a cigarette (usual brand or denicotinized depending on session and group). No cigarette will be smoked prior to fMRI-3. After smoking your cigarette you will sit in a quiet room and read magazines for 30 minutes. Following the 30 min rest period, you will be escorted to the fMRI suite at Duke University Medical Center. Once inside, you will complete questionnaires regarding your current mood and withdrawal symptoms. We will take a CO and saliva sample at the beginning of each scan. If you are wearing a nicotine replacement patch, you will remove it before entering the scanner. Then you will be given specific instructions regarding data collection procedures and be placed in the scanner. During the scanning you will perform each of the tasks, and lie still while we take pictures of your brain. After being removed from the scanner, you will complete post-session withdrawal and mood questionnaires and replace the removed patch. End-of-session instructions will then be provided:

* At the end of fMRI-1, ECIG participants will be released from the study. Smoker participants will be randomly assigned to either the EBT or NRT group, and given supplies and information regarding upcoming sessions.
* At the end of fMRI-2, you will be reminded of the quit date which you agreed upon previously, and you will be given supplies and information regarding quitting.
* At the end of fMRI-3, you will be given reminders about upcoming sessions.

You will be instructed not to consume any alcohol on the night before each scanning session.

We will ask for a breath and saliva sample before each session to make sure you have followed all directions about wearing the patch and smoking your usual brand or the denicotinized cigarettes as instructed. If the test indicates that you have not followed directions, you will be sent home (this will be considered a missed visit) and the visit will be re-scheduled. If this occurs on 2 consecutive visits, your further participation in the study will be terminated.

Follow-Up Sessions:

After completing all study visits, you will be asked to return for two follow-up sessions, one at 6 months and one at 12 months from visit 1. At these follow-up sessions we will ask for breath and saliva samples, and have you fill out paperwork regarding your mood and current smoking status.

ELIGIBILITY:
Inclusion Criteria (conventional cigarette smokers):

* generally healthy,
* between the ages of 18 and 55,
* smoking of at least 10 cigarettes/day of a brand delivering >0.5mg nicotine according to the standard Federal Trade Commission (FTC) method,
* an afternoon expired CO concentration of at least 10 ppm (to confirm inhalation),
* an interest in quitting smoking
* right-handed

Inclusion Criteria (e-cigarette smokers):

* generally healthy,
* between the ages of 18 and 55,
* prior history of smoking of at least 10 conventional cigarettes/day for at least two years of a brand delivering >0.5mg nicotine according to the standard Federal Trade Commission (FTC) method,
* no smoking of conventional cigarettes in the last 6 months;
* daily use of a nicotine-containing e-cigarette for at least 3 months;
* taking of at least 100 puffs per day from a nicotine-containing e-cigarette;
* an afternoon expired CO concentration <5 ppm (to confirm they are not combustible cigarette users);
* nicotine test strip reading >3
* right-handed

Exclusion Criteria:

* inability to attend all required experimental sessions,
* significant health problems (e.g., chronic hypertension (BP>150/90 sitting after 10 minutes), emphysema, seizure disorder, history of significant heart problems),
* use of psychoactive medications,
* use of smokeless tobacco,
* liver or kidney disorder (except kidney stones, gallstones)
* lung disorder (including but not limited to COPD, emphysema, and asthma)
* report of coronary heart disease; heart attack; cardiac rhythm disorder (irregular heart rhythm; chest pains; cardiac disorder (including but not limited to valvular heart disease, heart murmur, heart failure)
* current alcohol or drug abuse,
* use of illegal drugs as measured by urine drug screen,
* current use of nicotine replacement therapy or other smoking cessation treatment,
* presence of conditions that would make MRI unsafe (e.g., pacemaker, metal objects in the body, IUD, orthopedic pins or screws, etc.), or
* presence of conditions contraindicated for nicotine replacement therapy (e.g., skin allergies or disorders).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To test two quit smoking therapies and to study brain function while each therapy is being used. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States